CLINICAL TRIAL: NCT00453219
Title: Functional Hypothalamic Amenorrhea: Characterization of Metabolic Status, Brain Circuitry, and Stress-reactivity
Brief Title: FHA: Characterization of Metabolic Status, Brain Circuitry, and Stress-Reactivity
Status: Withdrawn | Type: Observational
Why Stopped: prior to participant recruitment, PI left Emory, study stopped
Sponsor: Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00024918
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Anovulation; FHA; Eumenorrhea; Polycystic Ovary Syndrome
MeSH Terms: conditions — Anovulation; Polycystic Ovary Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected, processed, and stored for the evaluation of genetic markers assocaited with stress vulnerability. Serum and plasma specimens will be collected and stored for the evaluation of factors associated with the regulation of reproduction.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Women ages 18-35 years with regular ovulatory menstrual cycles
  Interventions: Procedure: Screening evaluation; Procedure: Meal Response; Genetic: Blood Collection; Procedure: Functional MRI; Procedure: Endocrine Assessment
- 2: Women ages 18-35 years with irregular or absent menstrual periods due to functional hypothalamic amenorrhea (FHA) also called stress-induced anovulation
  Interventions: Procedure: Screening evaluation; Procedure: Meal Response; Genetic: Blood Collection; Procedure: Functional MRI; Procedure: Endocrine Assessment
- 3: Women ages 18-35 years with irregular or absent menstrual periods due to polycystic ovary syndrome(PCOS).
  Interventions: Procedure: Screening evaluation; Procedure: Meal Response; Genetic: Blood Collection; Procedure: Functional MRI; Procedure: Endocrine Assessment

INTERVENTIONS:
Procedure: Screening evaluation — A detailed history will be taken and a physical examination performed along with a blood sample to verify ovulatory status in women with regular cycles and determine cause of anovulation in women with irregular or absent menstrual cycles.
Procedure: Meal Response — The investigators are interested in how nutrition and metabolism can influence reproduction and they will look at how the body senses hunger and how it responses to food. Blood samples will be collected and questionnaires given to assess responses and feeling about hunger and food.
Genetic: Blood Collection — A blood sample will be collected and used to check for genetic markers of stress vulnerability.
Procedure: Functional MRI — research participants will have an functional MRI scan of their brain while reviewing word lists associated with body image and emotions. This procedure will last about 1 hour.
Procedure: Endocrine Assessment — research participants will have a 30 hour inpatient hospital admission with every 15 minute blood sampling for 24 hours. Hormone measures of stress, reproduction, and appetite will be obtained.

SUMMARY:
Functional Hypothalamic Amenorrhea (FHA), the spontaneous cessation of the menstrual cycle for at least 6 months after menstrual cyclicity has been established, is a common and reversible form of anovulation not due to discernible organic causes. Whereas animal studies suggest an interaction of metabolic and psychosocial stress in the genesis of FHA, the distinct central mechanisms in humans are not clear. On a behavioral level, FHA appears to depend on a complex interplay between individual stress susceptibility, stressful life events, and enduring metabolic challenge due to inappropriate attitudes towards eating and body image. We will use a comparison group of ovulatory, eumenorrheic women (EW) and a contrast group of lean women with polycystic ovary syndrome (PCOS). Although women with FHA and PCOS present with anovulation, each condition differs markedly in pathobiology (and health burden). Contrasting women with FHA to those with PCOS will afford an opportunity to understand more about the interaction between metabolism, stress, and reproduction and to determine the extent to which differences between FHA and EW are attributable to reproductive compromise (anovulation) per se versus specific to the pathogenesis of FHA or PCOS. We have used this approach to great advantage in the past to show that hypercortisolemia was confined to FHA and not PCOS (Berga 1997) and that dysfunctional (unrealistic) attitudes and decreased coping skills were reported more often in FHA than in PCOS and more in PCOS than EW. Further, this approach of comparing 3 groups will allow us to improve therapeutic approaches for two principle causes of anovulatory infertility in women. To accomplish this, we will study women with FHA, PCOS, and normal ovulatory women. The study will take place over 2 months and women will make 4-5 outpatient visits to the Clinical Integration Network Center and will have one overnight stay for frequent blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for participation are a gynecological age (age since menarche) > 5 and < 25 years, and chronological age > 18 years, within 90-110% of ideal body weight as determined by the 1983 Metropolitan height and weight table for women, and exercise < 10 h/wk and run < 10 mi/wk, day-awake/night-asleep schedule.
* Women in the FHA and PCOS groups have to fulfill the diagnostic criteria of FHA or PCOS and to have all other causes of amenorrhea and anovulation excluded.

Exclusion Criteria:

* Exclusion criteria are smoking, medications, including psychotropic or illicit drugs, medical, neurological, or ophthalmologic disease except acuity problems, a weight loss or gain of > 10 lb within a year preceding or since the onset of amenorrhea, a major Axis I disorder other than depression, parturition in the last 12 months and/or lactating in the last 6 months.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women ages 18-35
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-07

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Berga, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Background] Berga SL, Marcus MD, Loucks TL, Hlastala S, Ringham R, Krohn MA. Recovery of ovarian activity in women with functional hypothalamic amenorrhea who were treated with cognitive behavior therapy. Fertil Steril. 2003 Oct;80(4):976-81. doi: 10.1016/s0015-0282(03)01124-5. PMID 14556820
- [Background] Marcus MD, Loucks TL, Berga SL. Psychological correlates of functional hypothalamic amenorrhea. Fertil Steril. 2001 Aug;76(2):310-6. doi: 10.1016/s0015-0282(01)01921-5. PMID 11476778
- [Background] Berga SL, Loucks TL. Use of cognitive behavior therapy for functional hypothalamic amenorrhea. Ann N Y Acad Sci. 2006 Dec;1092:114-29. doi: 10.1196/annals.1365.010. PMID 17308138